CLINICAL TRIAL: NCT02973529
Title: Bioresorbable Vascular Stents for Treatment of Coronary Bifurcation Lesions Assessed by Optical Coherence Tomography - The BIFSORB Study
Brief Title: The Bioresorbable Implants for Scaffolding Obstructions in Randomized Bifurcations (BIFSORB) Study
Acronym: BIFSORB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, Principal investigator (MD, PhD), Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-215-14
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous intervention (PCI); Optical coherence tomography (OCT); Bifurcation lesion; Bioresorbable stents (BRS)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Absorb (Experimental): Randomization to implantation of Absorb BVS in bifurcation lesion
  Interventions: Device: Absorb
- Desolve (Experimental): Randomization to implantation of Desolve BRS in bifurcation lesion
  Interventions: Device: Desolve

INTERVENTIONS:
Device: Absorb — Randomization to implantation of Absorb BVS in bifurcation lesion
  Arms: Absorb
Device: Desolve — Randomization to implantation of Desolve BRS in bifurcation lesion
  Arms: Desolve

SUMMARY:
Coronary artery disease is often treated by implantation of permanent metallic stents.Coronary stents are required in the early healing phase after balloon dilatation but constitute a lifelong foreign body. New bioresorbable stents have been developed and are believed to improve long-term safety. The purpose of this study is to compare the safety and vessel healing after treatment of simple bifurcation lesions with the CE-marked bioresorbable stents Absorb and Desolve.

DETAILED DESCRIPTION:
BIFSORB is a prospective, randomized multicenter trial comparing 6-month healing outcome after treatment of simple coronary bifurcation lesions by Absorb or Desolve BRS. for treatment of coronary bifurcation lesions.

BRS are promising in treatment of coronary artery disease. The concept of bifurcation treatment using BRS is particular appealing as struts covering the side branch ostium may resorb over time.

The aim of this study is to compare the 6 months safety and vessel healing after treatment of coronary bifurcation lesions by the Desolve or Absorb BRS.

Hypothesis: Treatment of coronary bifurcation lesions using Absorb and Desolve bioresorbable stents is safe. Treatment of coronary bifurcation lesions by Desolve BRS is associated with a lower index of adverse vessel wall features (main vessel area stenosis, acquired malapposition, evaginations, late recoil, single end attached protruding struts, side branch ostial area stenosis) at 6 months compared to treatment with Absorb BRS.

Methods:

Prospective, open label, single blind, randomized, feasibility and safety pilot study with inclusion of 120 patients. Randomization 1:1 to Absorb or Desolve. Planned 6- and 24-month follow-up by OCT and follow-up for clinical endpoints until 10 years.

Eligible patients with a bifurcation lesion are treated by the provisional technique with mandatory jailing of the side branch and provisional opening of side branch ostium by the mini-kiss technique in case of severe pinching or TIMI-flow less than III. Proximal post-dilatation is mandatory. No dilatation beyond the expansion limits of the BRS.

The patients are assessed by optical coherence tomography (OCT) before, during and after implantation of the Absorb or Desolve BRS at baseline procedure and again at 6- and 24-month follow-up, or before if they are readmitted with a possible target lesion failure.

The operator is not blinded to pre-PCI OCT images that may be used for sizing and positioning of the scaffolds. Procedural OCT may be used to optimize scaffold implantation before performing final OCT.

Results are reported as clinical safety at 6 months (myocardial infarction, revascularization, death) and stent healing index by OCT including malapposition, stent coverage, side branch ostial area late loss, fracture and evaginations.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris
* Age > 18 years
* Stabilized non-ST elevation myocardial infarction
* Silent angina
* De novo coronary bifurcation lesions at LAD/diagonal, CX/obtuse marginal, RCA-PDA/posterolateral branch
* All Medina classes except Medina x.x.1
* Diameter of side branch ≥ 2.5 mm
* Signed informed consent

Exclusion Criteria:

* ST-elevation infarction within 48 hours
* Expected survival < 1 year
* Severe heart failure (NYHA≥III)
* S-creatinine > 120 µmol/L
* Allergy to contrast media, aspirin, clopidogrel, ticagrelor, ticlopidine, everolimus or novolimus
* Unable to cover main vessel lesion with one scaffold
* Severe tortuosity
* Severe calcification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-11 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Clinical safety measured as: major procedural myocardial infarction, non-procedural target vessel myocardial infarction, target lesion failure, cardiac death. | 6 months
  Clinical safety measured as: major procedural myocardial infarction, non-procedural target vessel myocardial infarction, target lesion failure, cardiac death.
Index of adverse vessel wall features | 6 months
  Side branch ostial area late loss, strut fracture, uncovered non-side branch apposed stent struts, uncovered stent struts in front of side branch, uncovered stent struts on acquired or persistent malapposed struts, persistent malapposition, max neointimal thickness/area stenosis, cumulated extra stent lumen gain

SECONDARY OUTCOMES:
Optical coherence tomography endpoint: acute malapposition | Baseline
Optical coherence tomography endpoint: acquired malapposition | 6 and 24 months
Optical coherence tomography endpoint: persistent malapposition | 6 and 24 months
Optical coherence tomography endpoint: Coverage of jailing struts | 6 and 24 months
Optical coherence tomography endpoint: Extra stent lumen (including evaginations) | Baseline, 6 and 24 months
Optical coherence tomography endpoint: Late stent recoil | 6 and 24 months
Optical coherence tomography endpoint: stent fracture | Baseline, 6 and 24 months
Optical coherence tomography endpoint: Single end attached protruding (floating) struts or neointimal tissue resembling struts | Baseline, 6 and 24 months
Optical coherence tomography endpoint: Ostial strut loss | Baseline, 6 and 24 months
Optical coherence tomography endpoint: Mean neointimal thickness | 6 and 24 months
Optical coherence tomography endpoint: Stent strut coverage | 6 and 24 months
Optical coherence tomography endpoint: Minimal luminal area in segmental analysis | Baseline, 6 and 24 months
Optical coherence tomography endpoint: Minimal stent area in segmental analysis | Baseline, 6 and 24 months
Optical coherence tomography endpoint: Minimum scaffold expansion area % | Baseline, 6 and 24 months
Optical coherence tomography endpoint: Segmental area stenosis | Baseline, 6 and 24 months
Optical coherence tomography endpoint: Healing above calcified plaque | 6 and 24 months
Optical coherence tomography endpoint: Healing above lipid plaque | 6 and 24 months
Optical coherence tomography endpoint: Acute thrombus on struts | Baseline
Optical coherence tomography endpoint: Late thrombus on struts | 6 and 24 months
Optical coherence tomography endpoint: Acute expansion | Baseline
  Measured in segments with; 1) calcified plaque, 2) lipid plaque, 3) area after predilatation < 30% of reference area, 4) stenosed segments (>50% area stenosis) with no dissections after predilatation
Optical coherence tomography endpoint:Late recoil | 6 and 24 months
  Measured in segments with; 1) calcified plaque, 2) lipid plaque, 3) area after predilatation < 30% of reference area, 4) stenosed segments (>50% area stenosis) with no dissections after predilatation
Angiographic endpoint: Ostial side branch area stenosis | Baseline, 6 and 24 months
Angiographic endpoint: Ostial side branch acute gain after main vessel stenting | Baseline
Angiographic endpoint: Ostial side branch late loss | 6 and 24 months
Angiographic endpoint: Ostial distal main vessel area stenosis | Baseline, 6 and 24 months
Angiographic endpoint: Ostial distal main vessel acute gain after main vessel stenting | Baseline
Angiographic endpoint: Ostial distal main vessel late loss | 6 and 24 months
Angiographic endpoint: Proximal main vessel area stenosis | Baseline, 6 and 24 months
Angiographic endpoint: Proximal main vessel acute gain after main vessel stenting | Baseline
Angiographic endpoint: Proximal main vessel late loss | 6 and 24 months
Angiographic endpoint: Minimal luminal area of all segments | Baseline, 6 and 24 months
Procedural endpoints: Procedure time | Baseline
  From sheath insertion to closure device excluding treatment of other vessels
Procedural endpoints: Contrast use | Baseline
Procedural endpoints: Fluoroscopy time | Baseline

OTHER OUTCOMES:
Clinical endpoints: Myocardial infarction | 10 years
Clinical endpoints: Target lesion failure | 10 years
Clinical endpoints: Target lesion revascularization | 10 years
Clinical endpoints: Stent thrombosis | 10 years
Clinical endpoints: Cardiac death | 10 years
Clinical endpoints: Non-Cardiac death | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Evald H Christiansen, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (4):
- Denmark (3):
  - Aarhus University Hospital, Aarhus N
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde, Roskilde
- Latvian Heart Center, Riga, Latvia

IPD SHARING:
Plan to Share IPD: Undecided